CLINICAL TRIAL: NCT01374347
Title: Brain SPECT Perfusion Imaging Following Cialis (Tadalafil ) Administration in Patients With Vascular Risk Factors
Brief Title: Brain SPECT Following Cialis (Tadalafil ) Administration
Acronym: CIALIS
Status: Completed | Type: Observational
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Mordechai Lorberboym Prof, PI, Wolfson Medical Center
Other Study IDs: 0044-11 WOMC
Record Dates: First submitted 2011-06-14; First posted 2011-06-15 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Change in Brain Perfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- One dose, Repeat doses: First group recives one dose Second group receives several doses
- One dose, several doses: 15 patients will take one dose of 20 mg cialis, and will have a second brain SPECT 24 hours after cialis administration. 15 other patients (age and risk factor matched) will be prescribed 5 mg of cialis once daily for 7 days, and a second SPECT study will be performed 24 hours after the last dose.

SUMMARY:
The study will be an open label one and will include 30 patients who underwent ischemic stroke 3 month to 3 years prior to the study. All patients will undergone a baseline brain SPECT perfusion study. 15 patients will take one dose of 20 mg cialis, and will have a second brain SPECT 24 hours after cialis administration. 15 other patients (age and risk factor matched) will be prescribed 5 mg of cialis once daily for 7 days, and a second SPECT study will be performed 24 hours after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients in the age range of 35-75 years.

Exclusion Criteria:

1. known allergic reaction to TF
2. Medical contraindication to use TF
3. Hemorrhagic stroke including intracerebral hemorrhage and subarachnoid hemorrhage
4. Acute stroke or cardiac ischemic event up to 3 month prior to study.
5. Other neurological brain diseases including degenerative diseases, multiple sclerosis, brain tumors, post severe brain injury (TBI) and migraine headache.
6. Sensory aphasia.
7. Cognitive impairment with disability to sign a consent form.Patients' Assessment

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients in the age range of 35-75 years.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)